CLINICAL TRIAL: NCT03329599
Title: Stroke Minimization Through Additive Anti-atherosclerotic Agents in Routine Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern California Institute of Research and Education (Other)
Collaborators: Kwame Nkrumah University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Bruce Ovbiagele, Chair, Neurology, Northern California Institute of Research and Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00068785
Record Dates: First submitted 2017-08-28; First posted 2017-11-06 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Atherosclerosis; Adherence, Medication; Tolerance
MeSH Terms: conditions — Atherosclerosis; Medication Adherence

STUDY DESIGN:
Intervention Model Description: SMAART incorporates (i) a pilot randomized controlled trial and (ii) a human capital/institutional capacity building component. We propose a randomized, open label, blinded endpoint clinical trial with the intervention arm assigned to a polypill containing 2/3 antihypertensives, a moderate/high-intensity statin and Aspirin to be taken orally, once daily in the form of a hard capsule compared with the 'usual care' arm who will continue to take separate, individual secondary preventive medications as prescribed their physicians to assess CIMT changes as a robust intermediary outcome measure for CVD events, as well as adherence, tolerability, and risk factor control rates. Furthermore, a cadre of emerging investigators from Ghana will benefit from the rich learning environment to be created through the implementation of the RCT and the interactions (2 years) with experts from the Medical University of South Carolina.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Polypill (Experimental): Assigned to a polypill containing 2/3 antihypertensives, a moderate/high-intensity statin and Aspirin to be taken orally, once daily in the form of a hard capsule
  Interventions: Drug: Polycap
- Usual Care (No Intervention): Will continue to take separate, individual secondary preventive medications as prescribed

INTERVENTIONS:
Drug: Polycap — Assigned to a polypill containing 2/3 antihypertensives, a moderate/high-intensity statin and Aspirin to be taken orally, once daily in the form of a hard capsule
  Arms: Polypill

SUMMARY:
The overarching objective of the Stroke Minimization through Additive Anti-atherosclerotic Agents in Routine Treatment (SMAART) trial is to assess whether a polypill containing fixed doses of (2/3) antihypertensives, a statin and antiplatelet therapy taken once daily orally would result in carotid intimal thickness regression-a surrogate marker of atherosclerosis, improved adherence, and tolerability compared with 'usual care' group on separate individual secondary preventive medications among Ghanaian first time stroke survivors. Our ultimate objective is to design of a future multi center, double-blinded, placebo-controlled, parallel-group, randomized trial comparing the clinical efficacy of the polypill strategy vs 'usual care' in the African context to derive locally relevant, high-quality evidence for routine deployment of polypill for CVD risk moderation among stroke survivors in LMICs. In this current study, we plan to recruit 120 recent ischemic stroke survivors randomized 1:1 to the polypill or usual care arms.

ELIGIBILITY:
Inclusion Criteria:

* Above the age of 18 years; male or female
* Stroke/TIA diagnosis no greater than two months before enrollment. Ischemic strokes including lacunar, large-vessel atherosclerotic, cardio-embolic subtypes are eligible -
* Subjects with stroke may present with at least one of the following additional conditions: Documented diabetes mellitus or previous treatment with oral hypoglycemic or insulin; documented hypertension >140/90mmHg or previous treatment with anti-hypertensive medications; Mild to moderate renal dysfunction (eGFR 60-30ml/min/1.73m2); Prior myocardial infarction
* Legally competent to sign informed consent

Exclusion Criteria:

* Unable to sign informed consent
* Contraindications to any of the components of the polypill
* Hemorrhagic stroke
* Severe cognitive impairment/dementia or severe global disability limiting the capacity of self-care
* Severe congestive cardiac failure (NYHA III-IV)
* Severe renal disease, eGFR <30ml/min/1.73m2), renal dialysis; awaiting renal transplant or transplant recipient
* Cancer diagnosis or treatment in past 2 years
* Need for oral anticoagulation at the time of randomization or planned in the future months
* Significant arrhythmias (including unresolved ventricular arrhythmias or atrial fibrillation)
* Nursing/pregnant mothers
* Do not agree to the filing, forwarding and use of his/her pseudonymized data.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenifer Voeks, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Kwame Nkrumah University of Science & Technology, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarfo FS, Adu-Gyamfi R, Opare-Addo PA, Agyei B, Ampofo M, Nguah SB, Ovbiagele B. Effect of a Cardiovascular Polypill on Poststroke Cognition Among Ghanaians: Secondary Analysis of a Randomized Clinical Trial. J Am Heart Assoc. 2024 Aug 6;13(15):e034346. doi: 10.1161/JAHA.124.034346. Epub 2024 Jul 31. PMID 39082406
- [Derived] Sarfo FS, Voeks J, Adamu S, Agyei BA, Agbenorku M, Adu-Darko N, Oteng MA, Obese V, Gyamfi RA, Mensah NA, Tagge R, Ampofo M, Kontoh SA, Nguah SB, Ovbiagele B. A cardiovascular polypill for secondary stroke prevention in a tertiary centre in Ghana (SMAART): a phase 2 randomised clinical trial. Lancet Glob Health. 2023 Oct;11(10):e1619-e1628. doi: 10.1016/S2214-109X(23)00347-9. PMID 37734804
- [Derived] Sarfo FS, Sarfo-Kantanka O, Adamu S, Obese V, Voeks J, Tagge R, Sethi V, Ovbiagele B. Stroke Minimization through Additive Anti-atherosclerotic Agents in Routine Treatment (SMAART): study protocol for a randomized controlled trial. Trials. 2018 Mar 14;19(1):181. doi: 10.1186/s13063-018-2564-0. PMID 29540234

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polypill | Usual Care
Started | 74 | 74
Completed | 59 | 64
Not Completed | 15 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polypill | Usual Care | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.7) | 58.1 (13.3) | 58.3 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 36 | 74
  Male | 36 | 38 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 74 | 74 | 148
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Ghana | 74 | 74 | 148
Educational Status [Count of Participants; unit: Participants]
  None | 11 | 15 | 26
  Primary | 42 | 28 | 70
  Secondary | 12 | 18 | 30
  Tertiary | 9 | 12 | 21
  Postgraduate | 0 | 1 | 1
Urban Residence [Count of Participants; unit: Participants] | 42 | 37 | 79
Marital Status [Count of Participants; unit: Participants]
  Never married | 6 | 5 | 11
  Married | 43 | 47 | 90
  Separated | 12 | 5 | 17
  Widow or widower | 11 | 14 | 25
  Cohabiting | 0 | 1 | 1
  Divorced | 2 | 2 | 4
Employment Status [Count of Participants; unit: Participants]
  Employed | 54 | 45 | 99
  Retired | 11 | 10 | 21
  Unemployed | 9 | 19 | 28
Monthly Income [Count of Participants; unit: Participants]
  0-100, US $ | 7 | 11 | 18
  101-250 | 37 | 37 | 74
  250-500 | 27 | 24 | 51
  >500 | 3 | 2 | 5
Hypertension [Count of Participants; unit: Participants] | 74 | 74 | 148
Haemoglobin A % [Mean (Standard Deviation); unit: percent] | 6.5 (1.7) | 7 (2.5) | 6.75 (2.14)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (4.3) | 25.7 (5.1) | 25.55 (4.72)
Waist-to-hip Ratio [Mean (Standard Deviation); unit: cm] | 92.2 (10.3) | 90.6 (12.1) | 91.4 (11.24)
Stroke subtype [Count of Participants; unit: Participants]
  Small vessel disease | 11 | 23 | 34
  Large vessel disease | 20 | 16 | 36
  Undetermined | 43 | 35 | 78
NIHSS Score [Mean (Standard Deviation); unit: score on a scale] — The NIH Stroke Scale/Score (NIHSS) quantifies stroke severity based on weighted evaluation findings.
  Ratings for each item are scored on a 3- to 5-point scale, with 0 as normal, and there is an allowance for untestable items. Scores range from 0 to 42, with higher scores indicating greater severity. Stroke severity may be stratified on the basis of NIHSS scores as follows: Very Severe: >25.
  score on a scale | 2.9 (3.4) | 2.4 (2.8) | 2.65 (2.66)
Modified Rankin Score [Mean (Standard Deviation); unit: score on a scale] — The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. 0 is the best score and 5 is the worst.
  score on a scale | 2.6 (0.97) | 2.74 (0.85) | 2.67 (0.91)
Common CIMT (Carotid Intima-Media Thickness) [Mean (Standard Deviation); unit: mm] | 1.00 (0.17) | 1.03 (0.16) | 1.02 (0.17)
Morisky Adherence Scale Score [Mean (Standard Deviation); unit: score on a scale] — The Morisky Medication Adherence Scale (MMAS-8) is a validated assessment tool used to measure non-adherence in a variety of patient populations. The scale has been verified and substantiated by numerous studies on a global scale with over 110 versions and over 80 translations.
  The MMAS-8 is an 8-item structured, self-report measure. Total scores on the MMAS-8 range from 0 to 8, with scores of:
  8 reflecting high adherence 7 or 6 reflecting medium adherence <6 reflecting low adherence
  0 is the worst score and 8 is the best.
  score on a scale | 6.7 (0.51) | 6.7 (0.37) | 6.7 (0.45)
Hill-Bone Score [Mean (Standard Deviation); unit: score on a scale] — The Hill-Bone Compliance to High Blood Pressure Therapy Scale is a 14-item scale that assesses patient behaviors for three important behavioral domains of high blood pressure treatment.
  (the three sub-scales of the original scale): Appointment Keeping (3-items), Diet (2-items), Medication Adherence (9-items).
  The scale has a four point response format: (4) all the time, (3) most of time, (2) some of time, and (1) never. Items are assumed to be additive, and, when summed, the total score ranges from 14 (minimum) to 56 (maximum). 14 is the worst and 56 is the best.
  score on a scale | 50.4 (1.81) | 50.1 (1.76) | 50.25 (1.79)
EQ-5D Quality-of-Life Score (Euro Quality of Life-5D) [Mean (Standard Deviation); unit: score on a scale] — The EQ-5D is a self-report survey that measures health-related quality of life. It consists of five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression.
  Each dimension has five response levels:
  No problems (Level 1) Slight Moderate Severe Extreme problems (Level 5)
  The EQ-5D also has a VAS scale from 0 (worst imaginable health state) to 100 (best imaginable health state). An individual records a score between 0 and 100 for their current overall health-related quality of life using the EQ VAS.
  score on a scale | 83.7 (11.6) | 80.6 (11.7) | 82.15 (11.65)
Treatment Satisfaction Questionnaire for Medication Score [Mean (Standard Deviation); unit: score on a scale] — The Treatment Satisfaction Questionnaire for Medication (TSQM) has scores that range from 0 to 100. Higher scores indicate higher patient satisfaction with medication. 0 is the worst, 100 is the best. The TSQM has 14 items and four domains:
  Effectiveness: Three items Side effects: Five items Convenience: Three items Global satisfaction: Three items The TSQM has a recall period of two to three weeks or since the last medication use. It was designed to assess patient treatment satisfaction in chronic diseases.
  score on a scale | 53.5 (2.8) | 52.7 (2.8) | 53.1 (2.8)
Montreal Cognitive Assessment Score [Mean (Standard Deviation); unit: score on a scale] — The Montreal Cognitive Assessment (MoCA) is a cognitive screening test that can detect dementia and mild cognitive impairment. The test consists of 11 questions that evaluate seven cognitive domains. The maximum score is 30.
  26 or higher: Normal 18-25: Mild cognitive impairment 10-17: Moderate impairment Less than 10: Severe impairment 0 is the worst, 30 is the best.
  score on a scale | 16.0 (6.7) | 16.2 (5.78) | 16.1 (6.26)
Hamilton Rating Scale for Depression Score [Mean (Standard Deviation); unit: score on a scale] — The Hamilton Rating Scale for Depression (HRSD) is a 21-item scale that is administered by a health care professional. The first 17 items are scored on either a 5-point or 3-point scale. The scale takes 15 to 20 minutes to complete and score.
  0-7: No depression 8-16: Mild depression 17-23: Moderate depression
  ≥24: Severe depression 0 is the best, 24 is the worst.
  score on a scale | 5.6 (4.36) | 6.8 (4.13) | 6.2 (4.25)
Systolic Blood Pressure, mmHg [Mean (Standard Deviation); unit: mmHg] | 161.3 (17.2) | 160.4 (18.0) | 160.85 (17.60)
Diastolic Blood Pressure, mmHg [Mean (Standard Deviation); unit: mmHg] | 92.0 (13.9) | 92.6 (14.6) | 92.3 (14.25)
Antiplatelet Therapy (aspirin or clopidogrel) [Count of Participants; unit: Participants] | 62 | 66 | 128
Atorvastatin at 40mg or 8mg daily [Count of Participants; unit: Participants] | 55 | 63 | 118
Angiotensin converting enzyme inhibitor [Count of Participants; unit: Participants] | 15 | 16 | 31
Angiotensin receptor blocker [Count of Participants; unit: Participants] | 43 | 43 | 86
Calcium channel blocker [Count of Participants; unit: Participants] | 62 | 58 | 120
Diuretics [Count of Participants; unit: Participants] | 25 | 29 | 54
Methyldopa [Count of Participants; unit: Participants] | 1 | 2 | 3
Hydralazine [Count of Participants; unit: Participants] | 10 | 8 | 18
Mineralocortcoid receptor blocker [Count of Participants; unit: Participants] | 7 | 7 | 14
β blocker [Count of Participants; unit: Participants] | 12 | 10 | 22
Diabetes [Count of Participants; unit: Participants] | 15 | 21 | 36
Cigarette Smoking [Count of Participants; unit: Participants] | 0 | 1 | 1
Alcohol use, current [Count of Participants; unit: Participants] | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Carotid Intimal Media Thickness
Description: Thickness of the intima and media layers of the carotid arteries
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Polypill | Usual Care
Number analyzed (Participants) | 59 | 64
mm | -0.017 [-0.067 to 0.034] | -0.092 [-0.130 to -0.051]

2. Secondary Outcome: Morisky Adherence Scale Score
Description: The Morisky Medication Adherence Scale (MMAS-8) is a validated assessment tool used to measure non-adherence in a variety of patient populations. The scale has been verified and substantiated by numerous studies on a global scale with over 110 versions and over 80 translations.
  The MMAS-8 is an 8-item structured, self-report measure. Total scores on the MMAS-8 range from 0 to 8, with scores of:
  8 reflecting high adherence 7 or 6 reflecting medium adherence <6 reflecting low adherence. 0 is the worst and 8 is the best.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Polypill | Usual Care
Number analyzed (Participants) | 59 | 64
score on a scale | -0.19 [-0.48 to 0.10] | -0.14 [-0.53 to 0.24]

3. Secondary Outcome: Hill-Bone Score
Description: The Hill-Bone Compliance to High Blood Pressure Therapy Scale is a 14-item scale that assesses patient behaviors for three important behavioral domains of high blood pressure treatment.
  (the three sub-scales of the original scale): Appointment Keeping (3-items), Diet (2-items), Medication Adherence (9-items).
  The scale has a four point response format: (4) all the time, (3) most of time, (2) some of time, and (1) never. Items are assumed to be additive, and, when summed, the total score ranges from 14 (minimum) to 56. 14 is the worst and 56 is the best.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Polypill | Usual Care
Number analyzed (Participants) | 59 | 64
score on a scale | -0.51 [-1.37 to 0.36] | -1.11 [-2.31 to 0.09]

4. Secondary Outcome: EQ-5D Quality-of-Life Score
Description: The EQ-5D is a self-report survey that measures health-related quality of life. It consists of five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression.
  Each dimension has five response levels:
  No problems (Level 1) Slight Moderate Severe Extreme problems (Level 5) The EQ-5D also has a VAS scale from 0 (worst imaginable health state) to 100 (best imaginable health state). An individual records a score between 0 and 100 for their current overall health-related quality of life using the EQ VAS.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Polypill | Usual Care
Number analyzed (Participants) | 59 | 64
score on a scale | 7.63 [5.08 to 10.18] | 10.23 [8.00 to 12.47]

5. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication Score
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) has scores that range from 0 to 100. Higher scores indicate higher patient satisfaction with medication. 0 is the worst, 100 is the best. The TSQM has 14 items and four domains:
  Effectiveness: Three items Side effects: Five items Convenience: Three items Global satisfaction: Three items The TSQM has a recall period of two to three weeks or since the last medication use. It was designed to assess patient treatment satisfaction in chronic diseases.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Polypill | Usual Care
Number analyzed (Participants) | 59 | 64
score on a scale | -10.92 [-15.88 to -5.96] | -6.72 [-10.80 to -2.63]

6. Secondary Outcome: Montreal Cognitive Assessment Score
Description: The Montreal Cognitive Assessment (MoCA) is a cognitive screening test that can detect dementia and mild cognitive impairment. The test consists of 11 questions that evaluate seven cognitive domains. The maximum score is 30.
  26 or higher: Normal 18-25: Mild cognitive impairment 10-17: Moderate impairment Less than 10: Severe impairment. 0 is the worst, 30 is the best.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Polypill | Usual Care
Number analyzed (Participants) | 59 | 64
score on a scale | 5.17 [4.17 to 6.17] | 5.39 [4.13 to 6.64]

7. Secondary Outcome: Modified Rankin Score
Description: The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is usually added for patients who expire. The Modified Rankin Score (mRS) is the most widely used outcome measure in stroke clinical trials. 0 is the best, 5 is the worst.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Polypill | Usual Care
Number analyzed (Participants) | 59 | 64
score on a scale | -0.92 [-1.14 to -0.69] | -0.89 [-1.09 to -0.69]

8. Secondary Outcome: Hamilton Rating Scale for Depression Score
Description: The Hamilton Rating Scale for Depression (HRSD) is a 21-item scale that is administered by a health care professional. The first 17 items are scored on either a 5-point or 3-point scale. The scale takes 15 to 20 minutes to complete and score.
  0-7: No depression 8-16: Mild depression 17-23: Moderate depression 0 is the best, 23 is the worst.
  ≥24: Severe depression
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Polypill | Usual Care
Number analyzed (Participants) | 59 | 64
score on a scale | -3.51 [-4.44 to -2.57] | -4.06 [-4.91 to -3.22]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Polypill | Usual Care
All-Cause Mortality (participants affected / at risk) | 5/74 | 2/74
Serious Adverse Events (participants affected / at risk) | 3/74 | 0/74
Other Adverse Events (participants affected / at risk) | 5/74 | 7/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Polypill (N=74) | Usual Care (N=74)
Post-stroke seizures (Vascular disorders) | 2 | 0
Hospitalization (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Polypill (N=74) | Usual Care (N=74)
Regimen Adjustments (Vascular disorders) | 5 | 7
Treatment Discontinuation (Vascular disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Gatrointestinal Bleeding (Gastrointestinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was conducted in a single tertiary medical centre, limiting its generalisability; The inter-rater agreement between the two independent CIMT readings per participants by the sonographers using a post-hoc intracluster correlation coefficient was fair; Future trials should be powered to assess treatment effects by stroke subtypes; Implementation of outcome measures must be performed to assess the barriers and facilitators associated with uptake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT03329599/Prot_SAP_000.pdf